CLINICAL TRIAL: NCT05193422
Title: Effects of Protective Face Masks on Cardiopulmonary Parameters at Rest and During Exercise in Children
Brief Title: Protective Face Masks and Cardiopulmonary Parameters at Rest and During Exercise in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Fouzas Sotirios, Assistant Professor of Pediatrics, University of Patras
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 10092020
Record Dates: First submitted 2021-11-03; First posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Face-masks; Exercise
Keywords: face-masks; exercise; children
MeSH Terms: conditions — Motor Activity | interventions — Oxygen Saturation; Heart Rate; Respiratory Rate; Temperature; Body Temperature; Humidity; Exercise Test

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to begin with Phase I followed by Phase II or Phase II followed by Phase I.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase I: No mask (Active Comparator): Participants, without wearing a face mask, will undergo the following:
  1. Measurement of peak nasal inspiratory flow
  2. Cardiopulmonary exercise testing (CPET) with an ergometric bike at 30% of their predicted maximum workload (Wmax) for 4 minutes, 50% of Wmax for 2 minutes and 70% of Wmax for 1 minute, with continuous oxygen saturation (SpΟ2), heart rate (HR), end-tidal CO2 (EtCO2) and respiratory rate (RR) monitoring.
  3. Spirometry and measurement of nPIF immediately after CPET.
  4. Discomfort assessment using a special scale
  Interventions: Diagnostic Test: Spirometry - baseline; Diagnostic Test: Spirometry - post CPET; Diagnostic Test: Nasal peak inspiratory flow - baseline; Diagnostic Test: Nasal peak inspiratory flow - post CPET; Diagnostic Test: Oxygen saturation; Diagnostic Test: Heart Rate; Diagnostic Test: End-tidal CO2; Diagnostic Test: Respiratory rate; Diagnostic Test: Cardiopulmonary exercise testing; Diagnostic Test: Discomfort level
- Phase II: Face mask (Experimental): Following nPIF measurement, participants will be asked to wear a standard surgical face mask. A temperature and humidity sensor will also be placed inside the mask. Will follow:
  1. Resting phase, 6 minutes. SpO2, HR, EtCO2 and RR will be monitored.
  2. CPET at 30% of Wmax for 4 minutes, 50% Wmax for 2 minutes and 70% Wmax for 1 minute. SpO2, HR, EtCO2 and RR will be continuously monitored.
  3. Spirometry and measurement of nPIF immediately after CPET.
  4. Discomfort assessment.
  Interventions: Diagnostic Test: Spirometry - post CPET; Diagnostic Test: Nasal peak inspiratory flow - baseline; Diagnostic Test: Nasal peak inspiratory flow - post CPET; Diagnostic Test: Oxygen saturation; Diagnostic Test: Heart Rate; Diagnostic Test: End-tidal CO2; Diagnostic Test: Respiratory rate; Diagnostic Test: Temperature; Diagnostic Test: Humidity; Diagnostic Test: Cardiopulmonary exercise testing; Diagnostic Test: Discomfort level

INTERVENTIONS:
Diagnostic Test: Spirometry - baseline — Standard spirometry using a Micro5000 spirometer to determine baseline FEV1, FVC, FEV1/FVC, FEF25-75 and PEF.
  Baseline spirometry will be performed before CPET in both study arms
  Arms: Phase I: No mask
Diagnostic Test: Spirometry - post CPET — Standard spirometry using a Micro5000 spirometer to determine baseline % change in FEV1 after CPET and assess exercise-induced bronchoconstriction (defined as FEV1 decrease >10% at 5 minutes after CPET) Post spirometry will be performed after CPET in both study arms
Diagnostic Test: Nasal peak inspiratory flow - baseline — Measurement of peak nasal inspiratory flow (nPIF) using a Micro5000 spirometer and a specially modified nasal mask.
  nPIF will be measured before CPET in both study arms
Diagnostic Test: Nasal peak inspiratory flow - post CPET — Measurement of peak nasal inspiratory flow (nPIF) using a Micro5000 spirometer and a specially modified nasal mask.
  nPIF will be measured after CPET in both study arms
Diagnostic Test: Oxygen saturation — Continuous monitoring of SpO2 using a Nonin 7500 pulse oximeter, in both study arms
  Other Names: SpO2
Diagnostic Test: Heart Rate — Continuous monitoring of HR using a Nonin 7500 pulse oximeter, in both study arms
  Other Names: HR
Diagnostic Test: End-tidal CO2 — Continuous monitoring of EtCO2 using a Microstream capnograph, in both study arms
  Other Names: EtCO2
Diagnostic Test: Respiratory rate — Continuous monitoring of RR using a Microstream capnograph, in both study arms
  Other Names: RR
Diagnostic Test: Temperature — Continuous monitoring of Temp in the face mask using a RHT03 sensor, only in the experimental study arm
  Other Names: Temp
  Arms: Phase II: Face mask
Diagnostic Test: Humidity — Continuous monitoring of Hum in the face mask using a RHT03 sensor, only in the experimental study arm
  Other Names: Hum
  Arms: Phase II: Face mask
Diagnostic Test: Cardiopulmonary exercise testing — CPET using an ULTIMA CPX device (MGC Diagnostics, Saint Paul, MI, USA) with an ergometric bike (eBike, GE Healthcare, Wauwatosa, WI, USA). Participants will be asked to exercise (steady pedaling at 60 rpm) at 30% of their predicted maximum workload (Wmax) for 4 minutes, at 50% of Wmax for 2 minutes and at 70% of Wmax for 1 minute. Wmax will be calculated as 3 Watts/kg.
  CPET will be performed in both study arms
  Other Names: CPET
Diagnostic Test: Discomfort level — Discomfort assessment using a special scale graded from 1 to 10 (Fikenzer, 2020).
  Both study arms, after CPET.

SUMMARY:
This study will examine the possible effects of protective surgical masks on the cardiorespiratory function of children aged 8-14 years at rest and during exercise.

The study will consist of two phases:

* Phase I: No face mask.

  1. Measurement of peak nasal inspiratory flow
  2. CPET with an ergometric bike at 30% of their predicted maximum workload (Wmax) for 4 minutes, 50% of Wmax for 2 minutes and 70% of Wmax for 1 minute, with continuous oxygen saturation (SpΟ2), heart rate (HR), end-tidal CO2 (EtCO2) and respiratory rate (RR) monitoring.
  3. Spirometry and measurement of nPIF immediately after CPET.
  4. Discomfort assessment using a special scale
* Phase II: Face mask. Following nPIF measurement, participants will be asked to wear a standard surgical face mask. A temperature and humidity sensor will also be placed inside the mask. Will follow:

  1. Resting phase, 6 minutes. SpO2, HR, EtCO2 and RR will be monitored.
  2. CPET at 30% of Wmax for 4 minutes, 50% Wmax for 2 minutes and 70% Wmax for 1 minute. SpO2, HR, EtCO2 and RR will be continuously monitored.
  3. Spirometry and measurement of nPIF immediately after CPET.
  4. Discomfort assessment.

Both phases will be performed on the same day with a recovery phase of 30 minutes between them. Participants will be randomized to begin with Phase I followed by Phase II or Phase II followed by Phase I.

At both phases, SpO2, HR, EtCO2 and RR (10 s average values) will be recorder at each 1 minute during CPET, and at minutes 0, 3 and 6 during the resting phase of Phase II. During Phase II, temperature and humidity will also be recorded at each 1 minute during CPET and at minutes 0, 3 and 6 during the resting phase.

The total duration of the protocol is estimated at 90 minutes per participant. The study sample will consist of 40 children stratified by age.

DETAILED DESCRIPTION:
PURPOSE

The purpose of this study is to investigate the possible effects of protective surgical masks on the cardiorespiratory function of children aged 8-14 years at rest and during exercise.

METHODS

A. Population

Children aged 8-14 years (minimum height 135 cm) will be invited to participate. They will be recruited from the outpatient clinics of the Pediatric Allergy and Pediatric Endocrinology Departments of the University Hospital of Patras, Greece. Children should not suffer from conditions that are likely to affect cardiopulmonary exercise testing (CPET) outcomes, such as respiratory (asthma and chronic lung disease), cardiac (congenital heart disease, heart failure), neurologic and musculoskeletal disorders.

The parents of the children will be informed about the aims of the study and they will be asked to give written consent. The study has been approved by the local Research and Ethics Committee (Act no. 407/9.10.2020).

B. Protocol

The study will be performed at the Respiratory Functions and CPET Laboratory of the Pediatric Pulmonary Unit. Children will present to the laboratory with one of their parents.

After history taking and measurement of weight and height, baseline spirometry will follow using a Micro5000 device (Medisoft, Sorinnes, Belgium) to determine FEV1, FVC, FEV1/FVC, FEF25-75 and PEF. The study will consist of two phases:

* Phase I: No face mask. Participants will perform

  1. Measurement of peak nasal inspiratory flow (nPIF) using the Micro5000 device and a specially modified nasal mask.
  2. CPET using an ULTIMA CPX device (MGC Diagnostics, Saint Paul, MI, USA) with an ergometric bike (eBike, GE Healthcare, Wauwatosa, WI, USA). Participants will be asked to exercise (steady pedaling at 60 rpm) at 30% of their predicted maximum workload (Wmax) for 4 minutes, at 50% of Wmax for 2 minutes and at 70% of Wmax for 1 minute. Wmax will be calculated as 3 Watts/kg.

     During CPET, oxygen saturation (SpΟ2) and heart rate (HR) will be continuously monitored using a Nonin 7500 pulse oximeter with a special ear sensor (Nonin Medical Inc, Plymouth, MN, USA). End-tidal CO2 (EtCO2) and respiratory rate (RR) will also be monitored using a Microstream device with special sampling (nasal) lines (Medtronic, Minneapolis, MN, USA).
  3. Spirometry and measurement of nPIF immediately after CPET.
  4. Discomfort assessment using a special scale graded from 1 to 10.
* Phase II: Face mask. Following nPIF measurement, participants will be asked to wear a standard surgical face mask. A temperature and humidity sensor (RHT03, MaxDetect Technologies, Shenzhen, China) will also be placed inside the mask on the right cheek, at nose level. Subsequently will follow:

  1. Resting phase, with the participants on the ergometric bike without pedaling and breathing normally for 6 minutes. SpO2, HR, EtCO2 and RR will be monitored during the resting phase.
  2. CPET at 30% of Wmax for 4 minutes, 50% of Wmax for 2 minutes and 70% of Wmax for 1 minute. SpO2, HR, EtCO2 and RR will be continuously monitored.
  3. Spirometry and measurement of nPIF immediately after CPET.
  4. Discomfort assessment.

Both phases will be performed on the same day with a recovery phase of 30 minutes between them. Participants will be randomized to begin with Phase I followed by Phase II or Phase II followed by Phase I.

At both phases, SpO2, HR, EtCO2 and RR (10 s average values) will be recorder at each 1 minute during CPET, and at minutes 0, 3 and 6 during the resting phase of Phase II. During Phase II, temperature and humidity will also be recorded at each 1 minute during CPET and at minutes 0, 3 and 6 during the resting phase.

The total duration of the protocol is estimated at 90 minutes per participant. The study sample will consist of 40 children stratified by age.

ELIGIBILITY:
Inclusion Criteria:

1. Children should not suffer from conditions that are likely to affect CPET outcomes, such as respiratory (asthma and chronic lung disease), cardiac (congenital heart disease, heart failure), neurologic and musculoskeletal disorders.
2. Height >135 cm
3. Parental written informed consent

Exclusion Criteria:

1. Points #1 or #2 not fulfilled
2. Child not willing to participate (e.g. not willing to wear the sensors)

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-01-20 (Estimated); Primary Completion 2022-02-20 (Estimated); Study Completion 2022-03-20 (Estimated)

PRIMARY OUTCOMES:
SpO2 | Minute 1
  Oxygen saturation
SpO2 | Minute 2
  Oxygen saturation
SpO2 | Minute 3
  Oxygen saturation
SpO2 | Minute 4
  Oxygen saturation
SpO2 | Minute 5
  Oxygen saturation
SpO2 | Minute 6
  Oxygen saturation
SpO2 | Minute 7
  Oxygen saturation
HR | Minute 1
  Heart rate
HR | Minute 2
  Heart rate
HR | Minute 3
  Heart rate
HR | Minute 4
  Heart rate
HR | Minute 5
  Heart rate
HR | Minute 6
  Heart rate
HR | Minute 7
  Heart rate
EtCO2 | Minute 1
  End-tidal CO2
EtCO2 | Minute 2
  End-tidal CO2
EtCO2 | Minute 3
  End-tidal CO2
EtCO2 | Minute 4
  End-tidal CO2
EtCO2 | Minute 5
  End-tidal CO2
EtCO2 | Minute 6
  End-tidal CO2
EtCO2 | Minute 7
  End-tidal CO2
RR | Minute 1
  Respiratory rate
RR | Minute 2
  Respiratory rate
RR | Minute 3
  Respiratory rate
RR | Minute 4
  Respiratory rate
RR | Minute 5
  Respiratory rate
RR | Minute 6
  Respiratory rate
RR | Minute 7
  Respiratory rate
Temperature | Minute 1
  Air temperature (in degrees Celsius) within the face mask
Temperature | Minute 2
  Air temperature (in degrees Celsius) within the face mask
Temperature | Minute 3
  Air temperature (in degrees Celsius) within the face mask
Temperature | Minutε 4
  Air temperature (in degrees Celsius) within the face mask
Temperature | Minute 5
  Air temperature (in degrees Celsius) within the face mask
Temperature | Minute 6
  Air temperature (in degrees Celsius) within the face mask
Temperature | Minute 7
  Air temperature (in degrees Celsius) within the face mask
Humidity | Minute 1
  Relative air humidity (%) within the face mask
Humidity | Minute 2
  Relative air humidity (%) within the face mask
Humidity | Minute 3
  Relative air humidity (%) within the face mask
Humidity | Minute 4
  Relative air humidity (%) within the face mask
Humidity | Minute 5
  Relative air humidity (%) within the face mask
Humidity | Minute 6
  Relative air humidity (%) within the face mask
Humidity | Minute 7
  Relative air humidity (%) within the face mask
Discomfort level | Minute 7
  Level of discomfort (specific questionnaire (5 items), scale 1 to 10) after CPET
Exercise-induced bronchoconstriction | Minute 7
  % change in FEV1 value before-after CPET
% change in nPIF | Minute 7
  % change in nPIF value before-after CPET

CONTACTS AND LOCATIONS:
Overall Officials: Sotirios Fouzas, Prof., Principal Investigator — Pediatric Respiratory Unit, University Hospital of Patras, Greece; Michael Anthracopoulos, Prof., Study Chair — Pediatric Respiratory Unit, University Hospital of Patras, Greece